CLINICAL TRIAL: NCT05269446
Title: Total-body 18F-PBR06 PET/CT to Evaluate Systemic Inflammation and Perfusion in STEMI and SA Patients Receiving PCI
Brief Title: 18F-PBR06/Total Body PET Imaging in Patients With STEMI
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: STEMI-systemic inflammation
Record Dates: First submitted 2022-01-05; First posted 2022-03-08 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected at D7 and D180 after enrolment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- STEMI patients: STEMI: patients diagnosed with ST-segment elevation myocardial infarction
  Interventions: Procedure: percutaneous coronary intervention (PCI); Device: total body PET/CT scan; Procedure: Coronary Angiography (CAG); Drug: TSPO injection
- SA or NSTEMI patients: SA: patients diagnosed with stable angina
  Interventions: Procedure: percutaneous coronary intervention (PCI); Device: total body PET/CT scan; Procedure: Coronary Angiography (CAG); Drug: TSPO injection
- Healthy subjects: Patients with suspected coronary artery disease, but coronary angiography (CAG) indicates no obvious coronary stenosis
  Interventions: Device: total body PET/CT scan; Procedure: Coronary Angiography (CAG); Drug: TSPO injection

INTERVENTIONS:
Procedure: percutaneous coronary intervention (PCI) — A family of minimally invasive procedures used to open clogged coronary arteries and restore blood flow. This is also a standard treatment for patients diagnosed with STEMI or SA
  Groups: SA or NSTEMI patients; STEMI patients
Device: total body PET/CT scan — all participants will receive a total-body PET/CT scan (uExplorer) after enrolment
Procedure: Coronary Angiography (CAG) — A procedure that uses X-ray imaging to visualize coronary arteries.
Drug: TSPO injection — Participants will receive one dose of the non-therapeutic administration of the radioactive TSPO tracer 18F-PBR06 before a whole-body scan by uExplorer

SUMMARY:
The study will use 18F-PBR06/uExplorer to study the activation of macrophages and systemic perfusion in patients with ST-segment elevation myocardial infarction (STEMI) or stable angina (SA). Participants will receive the total-body PET/CT scan on the seventh day (Day 7, D7) and D180 of enrolment.

DETAILED DESCRIPTION:
The aim of our study is to explore the activation of macrophages in patients with ST-segment elevation myocardial infarction (STEMI) or stable angina (SA) using the 18 kDa translocator protein (TSPO) radioligand 18F N-fluoroacetyl-N-(2,5-dimethoxybenzyl)-2-phenoxyaniline (18F-PBR06) in combination with the world's first commercially available total-body PET/CT (uExplorer). The investigators expect to enroll 10 patients diagnosed with STEMI and 10 patients with SA who receive coronary angiography (CAG) and the percutaneous coronary intervention (PCI), and 5-10 healthy individuals diagnosed with SA but presenting negative CAG at Renji Hospital, Shanghai. The activation of macrophages (TSPO uptake) and blood perfusion in different organs will be studied using 18F-PBR06/uExplorer.

With written consent from eligible participants, the investigators will review past medical records and document the medical history for each participant. Patients will undergo PCI on the day of enrolment (12 hours within the symptom onset for STEMI patients). Screen procedures will be performed at the seventh day of enrolment (Day 7, D7) and Day 180 (D180). Participants will receive one dose of the non-therapeutic administration of the radioactive TSPO tracer 18F-PBR06 and receive a whole-body scan by uExplorer. TSPO uptake and blood flow in the heart, kidney, liver, brain, and lung will be recorded. All participants will be followed for 1 year after enrolment. Blood samples will be collected and echocardiography will be performed at D7 and D180. Major adverse cardiovascular events (MACE) will be recorded throughout the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years old
* Diagnosed with STEMI, NSTEMI or suspected SA (ACC/AHA guidelines)
* Half male and half female
* Undergo CAG and PCI treatment if necessary (primary PCI for STEMI patients within12 hours after symptom onset)
* Written informed consents will be offered and signed by all participants

Exclusion Criteria:

* History of myocardial infarction/vascular disease/heart failure/systemic inflammatory diseases before enrolment
* Patients who are pregnant/breastfeeding, or in a plan to have a baby during the year after CAG/PCI
* People under the age of 18 years old
* Inability to lie or maintain posture during the scanning procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — half male and half female
Study Population: Patients aged between 18 and 75 years with the diagnosis of STEMI or SA will be eligible for our study.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-11-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline TSPO uptake (SUV max) at 6 month | Day 7 and Day 180 after enrolment
  TSPO uptake is assessed by drawing regions of interest (ROI), and determined as the mean of maximal standard uptake value (SUV max)
Change from baseline Blood flow value (ml/g/min) at 6 month | Day 7 and Day 180 after enrolment
  Blood flow value is quantified using a reconstructed model, and determined as ml/g/min

SECONDARY OUTCOMES:
Incidence of MACE (%)in patients with STEMI and SA | Throughout the 1 year follow-up
  The rate of patients with major adverse cardiovascular events (MACE) occurring during the follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No